CLINICAL TRIAL: NCT01749423
Title: A Retrospective Study to Evaluate the Effectiveness of onabotulinumtoxinA in Preventing Headaches in Patients With Chronic Migraines
Status: Withdrawn | Type: Observational
Why Stopped: Company decision due to enrollment challenges.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTX-CM-12-518
Record Dates: First submitted 2012-12-12; First posted 2012-12-13 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Previous treatment with onabotulinumtoxinA for Chronic Migraine based on retrospective review of medical records.
  Interventions: Biological: OnabotulinumtoxinA

INTERVENTIONS:
Biological: OnabotulinumtoxinA — Previous treatment with onabotulinumtoxinA for Chronic Migraine.
  Other Names: botulinum toxin Type A; BOTOX®

SUMMARY:
This study will evaluate the effectiveness of OnabotulinumtoxinA to prevent headaches in patients with Chronic Migraine.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic migraines
* 15 or more headache days over a 30 day period
* A minimum of 2 consecutive treatment cycles of 100 units onabotulinumtoxinA and a minimum of 2 consecutive treatment cycles with the onabotulinumtoxinA dosing between 155 and 195 units

Exclusion Criteria:

* Any treatment cycle dose of onabotulinumtoxinA greater than 200 units

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic migraines who received a minimum of two consecutive treatment cycles of 100 units onabotulinumtoxinA and a minimum of two consecutive treatment cycles with the OnabotulinumtoxinA dosing between 155 and 195 units.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of Headache Days | Up to 56 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan